CLINICAL TRIAL: NCT02804230
Title: A Feasibility Study to Evaluate Safety and Initial Effectiveness of MR-Guided Focused Ultrasound Ablation Therapy in the Treatment of Focal Epilepsy
Brief Title: MR-Guided Focused Ultrasound in the Treatment of Focal Epilepsy (EP001)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: InSightec (Industry)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP001
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy
Keywords: Mr-Guided Focused Ultrasound
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, single-cohort study with no control group to evaluate initial safety, feasibility, and effectiveness of the Exablate 4000 Type 1 or 1.1 System.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (1):
- Exablate Neuro System Treatment (Experimental): MR-Guided Focused Ultrasound will be used to ablate epileptic foci up to 8 cm3 in size.
  Interventions: Device: Neuro Ablation - Functional

INTERVENTIONS:
Device: Neuro Ablation - Functional — MR-Guided Focused Ultrasound
  Other Names: Focused Ultrasound; MRgFUS; FUS

SUMMARY:
The purpose of this study is to evaluate the feasibility, safety, and initial effectiveness of Exablate thermal ablation of a focal epileptic target area in the brain of patients suffering from medication-refractory epilepsy, using the Exablate transcranial system to produce multiple sonications targeted in the focus of interest. The investigators will establish the feasibility and collect data to establish the basic safety of this type of treatment as the basis for later studies that will evaluate its full clinical efficacy.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the feasibility, safety, and initial effectiveness of Exablate thermal ablation of a focal epileptic target area in the brain of patients suffering from medication-refractory epilepsy, using the Exablate transcranial system to produce multiple sonications targeted in the lesion of interest. The Investigators will establish the feasibility and collect data to establish the basic safety of this type of treatment as the basis for later studies that will evaluate its full clinical efficacy.

The hypotheses tested are that:

1. MRgFUS treatment of focal epilepsy is feasible and safe, with a low risk of adverse effects as evaluated during the follow-up period.
2. Exablate treatment of foci in patients with focal epilepsy reduces the seizure frequency.

ELIGIBILITY:
Inclusion Criteria:

Patients who are able and willing to give consent and able to attend all study visits.

Seizure refractory to at least three standard antiepileptic medications at adequate doses, failed for lack of efficacy. This may include a rescue medication designated use as PRN.

A minimum of 3 seizures per month for 2 months by patient diary started at intake interview.

Subjects should have focal seizures with or without secondary generalization. Subjects should have evidence suggesting the focus within the periventricular white matter, basal ganglia, thalamus, hypothalamus, or mesial temporal lobe has been previously determined as the source of seizures by standard clinical criteria including at least the description of seizures, physical examination, neuroimaging, and video EEG monitoring capturing at least one seizure.

Subjects must be taking 2 medications during the Baseline period and the dosage must be stable.

A diagnosis of intractable lesional epilepsy which may include: Hypothalamic hamartoma, Periventricular nodular hetereotopia, Dysembryoplastic neuroepithelial tumor (DNET), Cortical dysplasia, Tuberous sclerosis, Focal cortical gliosis, or Predominately unilateral Mesial Temporal Lobe Epilepsy (MTLE).

Exclusion Criteria:

Patients with unstable cardiac status that would increase anesthetic risk including: unstable angina pectoris on medication, documented myocardial infarction within six months of protocol entry, congestive heart failure requiring medication (other than diuretic), anti-arrhythmic drug use.

Patients exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV as manifested by one (or more) of the following occurring within a 12 month period:

Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (such as repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; or neglect of children or household, Recurrent substance use in situations in which it is physically hazardous (such as driving an automobile or operating a machine when impaired by substance use), Recurrent substance-related legal problems (such as arrests for substance related disorderly conduct), Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (for example, arguments with spouse about consequences of intoxication and physical fights).

Severe hypertension (diastolic BP > 100 on medication) measured at intake interview or on Treatment Day.

Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.

Known intolerance or allergies to the MRI contrast agent (i.e. Gadavist) including advanced kidney disease.

Known or suspected sensitivity to perfluetren (Definity®). Severely impaired renal function (estimated glomerular filtration rate < 45ml/min/1.73 m2) or receiving dialysis.

History of abnormal bleeding and/or coagulopathy. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk of hemorrage (e.g. Avastin) within one month of focused ultrasound procedure; or, unable or unwilling to stop anticoagulant for the purposed of focused ultrasound procedure.

Active or suspected acute or chronic uncontrolled infection. History of intracranial hemorrhage. Cerebrovascular disease (multiple CVA or CVA within 6 months). Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hrs of total table time).

Symptoms and signs of increased intracranial pressure (e.g. headache, nausea, vomiting, lethargy, and papilledema).

Are participating or have participated in another clinical trial in the last 30 days.

Presence of any other neurodegenerative disease. Present of cognitive impairment severe enough to be unable to understand and consent for the study, or understand the procedures.

History of immunocompromise, including patient who is HIV positive. Known life-threatening systemic disease. Patient with current or a prior history of current suicidal ideation or previous suicide attempt within the past year.

Patients with risk factors for intraoperative or postoperative bleeding (platelet count less than 100,000 per cubic millimeter, PT > 14, PTT > 36 or INR > 1.3) or a documented coagulopathy.

Patients with malignant brain tumors. Any illness that in the investigator's opinion precludes participation in this study.

Pregnancy or lactation. Legal incapacity or limited legal capacity. Patients with a known history of psychogenic non-epileptic spells in the last three years.

Patients with a vagal nerve stimulator (that is not MRI-safe and/or MRI compatible), deep brain stimulator, other implanted electronic device, or prior radiofrequency lesion techniques.

Patient with cardiopulmonary or vascular illness that would complicate anesthesia.

Patients who are unwilling to undergo general anesthesia. Patients with lesions in the brainstem or cerebellum. Patients with symptomatic generalized epilepsy. Patients with only simple partial seizures. Patients who have had convulsive status epilepticus within 12 months prior to baseline.

Patients with a prior diagnosis of psychogenic/non-epileptic seizures within the last 5 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06-07 (Actual); Primary Completion 2023-06-23 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of device and procedure related complications | At the time of Exablate transcranial procedure

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - University of Virginia, Charlottesville, Virginia